CLINICAL TRIAL: NCT00448565
Title: Prediction of Extubation Success by the Patient
Status: Completed | Type: Observational
Sponsor: Ospedale Regionale Bellinzona e Valli (Other)
Responsible Party: Ospedale Regionale Bellinzona e Valli, ICU
Other Study IDs: CEC-06-2807
Record Dates: First submitted 2007-03-15; First posted 2007-03-19 (Estimated); Last update posted 2009-02-02 (Estimated); Status verified 2009-01

CONDITIONS: Mechanical Ventilation; Respiratory Failure; Extubation
Keywords: extubation; prediction
MeSH Terms: conditions — Respiratory Insufficiency

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

SUMMARY:
The evidence-based approach to wean and consecutively extubate patients is based solely on objective criteria/tests. The introduction of subjective criteria could further improve the actual method.

ELIGIBILITY:
Inclusion Criteria:

* all intubated patients ready for a spontaneous breathing trial

Exclusion Criteria:

* not awake
* not collaborative

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients in interdisciplinary ICU
Sampling Method: Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2007-01

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Perren, MD, Principal Investigator — Ospedale Regionale Bellinzona e Valli
Locations (2):
- Switzerland (2):
  - Ospedale Regionale Bellinzona e Valli, Bellinzona, Canton Ticino
  - University hospital, Service des Soins intensifs, Geneva